CLINICAL TRIAL: NCT06693050
Title: AQT90 FLEX NTproBNP2 Test Kit Method Comparison Study
Status: Completed | Type: Observational
Sponsor: Radiometer Medical ApS (Industry)
Responsible Party: Sponsor
Other Study IDs: DC-087457
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Diagnostic Test

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to verify performance claims for method comparison for the NTproBNP2 Test Kit on the AQT90 FLEX analyzer in whole blood (WB) and plasma (PL).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able to understand given information and demonstrate willingness and ability to voluntarily give a signed, valid written informed consent to participate in the study.
* Subjects must be 18 years of age or older.
* Subjects with expected NT-proBNP concentrations within the measuring range of NTproBNP2 assay.

Exclusion Criteria:

* Subjects known to be pregnant or breast-feeding.
* Subjects previously enrolled in the study.
* Subject, who has withdrawn consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient population with expected NT-proBNP concentrations within the measuring range of NTproBNP2 assay.
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2024-12-09 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
Slope, R | 5 month
  Slope, R, for NTproBNP2 Test Kit on the AQT90 FLEX analyzer vs. Elecsys proBNP II assay across sites

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Hospiltal Universitari Germans Trias i Pujol, Badalona
  - Clinica Universidad de Navarra, Madrid
  - Servicio Andaluz de Salud (SAS) - Hospital San Juan de la Cruz, Ùbeda